CLINICAL TRIAL: NCT06345963
Title: Enhancing Brain Connectivity in Schizophrenia Through Neuromodulation (Study 1)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Xiaoming Du, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-23-1044 (study 1)
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Schizophrenia
Keywords: Transcranial magnetic stimulation; schizophrenia; white matter; connectivity; myelination
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active rTMS (Experimental): Participants in this group will receive active H-coil delivered rTMS.
  Interventions: Device: active H-coil delivered rTMS

INTERVENTIONS:
Device: active H-coil delivered rTMS — Multiple trains of rTMS in a day, for multiple days.

SUMMARY:
Patients with schizophrenia spectrum disorder (SSD) will be exposed to active repetitive transcranial magnetic stimulation (rTMS) from H coil for improving white matter integrity.

DETAILED DESCRIPTION:
Schizophrenia is a severe mental illness that affects about 1% of the population but a major source of disability. Information processing between brain regions occurs due to transfer of electrical impulses among them. This process is determined by the existing neuronal/fiber connections, which may be altered and or modified in the presence of neuronal stimulation or cognitive intervention. The frontal lobe information flow is critical for higher cognitive functions, thought processes, and proper emotional and behavioral responses. Improving the myelination in the frontal lobe may increase cognitive functions and reduce risks to develop symptoms of schizophrenia. The investigators propose that increasing electrical signaling in the frontal white matter in patients with schizophrenia may also enhance myelination and improve the white matter integrity.

The patients with schizophrenia will receive active repetitive transcranial magnetic stimulation (rTMS) treatment. The rTMS with H coil is FDA-cleared for short-term smoking cessation in the general population. Its efficacy in myelination modulation has not been evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female ages between ages 18-60 years
2. Ability to give written informed consent (age 18 or above)
3. Diagnosed with schizophrenia-spectrum disorder and Evaluation to Sign Consent (ESC) above 10.

Exclusion Criteria:

1. Inability to sign informed consent.
2. Any history of seizures.
3. Any acute and unstable major medical illnesses that may affect normal brain functioning. Examples of these conditions include, but not limited to, recent stroke, seizure, history of significant head trauma, CNS infection or tumor, other significant brain neurological conditions (As this is a study of medical comorbidity, most medical conditions, once stable, are not exclusion criteria).
4. Taking > 400 mg clozapine/day.
5. Failed TMS screening questionnaire.
6. Significant alcohol or other drug use (substance dependence within 6 months or substance abuse within 1 month) other than nicotine or marijuana dependence.
7. A history of thrombosis, family history of thrombosis, or medical conditions that may lead to a hypercoagulable state (increased chance to develop blood clots)
8. Woman who is pregnant (child-bearing potential but not on contraceptive and missing menstrual period; or by self-report; or by positive urine pregnancy test).
9. History of head injury with loss of consciousness over 10 minutes; history of brain surgery
10. Cannot refrain from using alcohol and/or marijuana 24 hours or more prior to experiments.
11. Students and employees currently involved with our lab (lab employees and personnel will be excluded from the study to avoid possible coercion or possible appearance of coercion, or chance of breach of privacy and confidentiality).
12. For MRI, unable to undergo MRI scanning due to metallic devices or objects (cardiac pacemaker or neurostimulator, some artificial joints, metal pins, surgical clips, or other implanted metal parts) or claustrophobic to the scanner.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2029-05-01 (Estimated); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Brain microstructural integrity as indicated by white matter fractional anisotropy (FA) values as assessed by magnetic resonance imaging (MRI) | baseline, visit 6 (about 1 week after baseline), visit 10 (about 2 weeks after baseline)
  Fractional anisotropy (FA) values will be reported. FA values range from 0 to 1 with larger values indicating greater white matter integrity.
Brain connectivity as indicated by resting-state functional connectivity (rsFC) values as assessed by functional MRI (fMRI) | baseline, visit 6 (about 1 week after baseline), visit 10 (about 2 weeks after baseline)
  rsFC values will be reported as a Z-score with a range of -1 to 1, with greater absolute values indicating stronger brain connectivity.

SECONDARY OUTCOMES:
Electrophysiological response as indicated by mismatch negativity as assessed by electroencephalography (EEG) | baseline, visit 6 (about 1 week after baseline), visit 10 (about 2 weeks after baseline)
  Mismatch negativity values will be reported in microvolts (uV). Mismatch negativity is measured by subtracting the averaged response to a set of standard stimuli from the average response to deviant stimuli, and taking the amplitude of this difference in a given timepoint.
Electrophysiological response as indicated by steady-state auditory evoked responses from electroencephalography recording (EEG) | baseline, visit 6 (about 1 week after baseline), visit 10 (about 2 weeks after baseline)
  Steady-state auditory evoked responses will be reported. The responses are measured by calculating the ratio of the power at target frequency over power at the surrounding background frequencies. The ration will be obtained in a given timepoint.
Cognitive insight as assessed by the Beck Cognitive Insight Scale | baseline, visit 6 (about 1 week after baseline), visit 10 (about 2 weeks after baseline)
  Total score will be reported and ranges from 15 to 60, with a higher score indicating greater cognitive insight.
Depression as assessed by the Depression State and Trait Scale (DST) - state | baseline, visit 6 (about 1 week after baseline), visit 10 (about 2 weeks after baseline)
  Total score of the state subscale of the DST will be reported and ranges from 0 to 72, with a higher score indicating greater depression state.
Depression as assessed by the Depression State and Trait Scale (DST) - trait | baseline, visit 6 (about 1 week after baseline), visit 10 (about 2 weeks after baseline)
  Total score of the trait subscale of the DST will be reported and ranges from 0 to 72, with a higher score indicating greater depression trait.
Depression as assessed by the Calgary Depression Scale | baseline, visit 6 (about 1 week after baseline), visit 10 (about 2 weeks after baseline)
  Total score of the Calgary Depression Scale will be reported and ranges from 0 to 27, with a higher score indicating greater depression.
Depression as assessed by the Beck Depression Inventory | baseline, visit 6 (about 1 week after baseline), visit 10 (about 2 weeks after baseline)
  Total score of the Beck Depression Inventory will be reported and ranges from 0 to 63, with a higher score indicating greater depression.
Perception as assessed by the Perception State and Trait Scale - state | baseline, visit 6 (about 1 week after baseline), visit 10 (about 2 weeks after baseline)
  The Perception State and Trait Scale assesses alterations in the perception of audio and visual experiences. Total score ranges from 0 to 96 for the state subscale, and a higher score indicates a greater alteration of audio or visual experiences state.
Perception as assessed by the Perception State and Trait Scale - trait | baseline, visit 6 (about 1 week after baseline), visit 10 (about 2 weeks after baseline)
  The Perception State and Trait Scale assesses alterations in the perception of audio and visual experiences. Total score ranges from 0 to 96 for the trait subscale, and a higher score indicates a greater alteration of audio or visual experiences trait.
Delusion as assessed by the 21-item Peters Delusion Inventory (PDI-21) | baseline, visit 6 (about 1 week after baseline), visit 10 (about 2 weeks after baseline)
  Total score will be reported and ranges from 0 to 21, with a higher score indicating greater delusion.
Emotion regulation as assessed by the Profile of Mood States (POMS) | day 1 after baseline, day 2 after baseline, day 3 after baseline, day 4 after baseline, day 5 after baseline, day 9 after baseline, day 10 after baseline
  Total score will be reported and ranges from 0 to 204, with a higher score indicating more positive emotion and mood. This outcome measure will be assessed at each of the 10 treatment visits (which are about day 1 after baseline, day 2 after baseline, day 3 after baseline, day 4 after baseline, day 5 after baseline, day 9 after baseline, day 10 after baseline, respectively).
Hallucination as assessed by the Revised Hallucinations Scale (RHS) | day 1 after baseline, day 2 after baseline, day 3 after baseline, day 4 after baseline, day 5 after baseline, day 9 after baseline, day 10 after baseline
  Total score will be reported and ranges from 0 to 13, with a higher score indicating greater hallucination. This outcome measure will be assessed at each of the 10 treatment visits (which are about day 1 after baseline, day 2 after baseline, day 3 after baseline, day 4 after baseline, day 5 after baseline, day 9 after baseline, day 10 after baseline, respectively).
Cognitive function as assessed by the Letter-Number Span subscale of the MATRICS consensus cognitive battery (MCCB) | baseline, visit 6 (about 1 week after baseline), visit 10 (about 2 weeks after baseline)
  Total score will be reported and ranges from 0 to 24, with a higher score indicating greater cognitive function.
Cognitive function as assessed by the Spatial Span subscale of the MATRICS consensus cognitive battery (MCCB) | baseline, visit 6 (about 1 week after baseline), visit 10 (about 2 weeks after baseline)
  Total score will be reported and ranges from 0 to 32, with a higher score indicating greater cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoming Du, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center, Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No